CLINICAL TRIAL: NCT03857048
Title: Adaptive Responses to Overfeeding and Weight Regain in Reduced Obese Individuals
Brief Title: Adaptive Responses to Overfeeding and Weight
Acronym: ARrOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-0091
Record Dates: First submitted 2018-10-22; First posted 2019-02-27 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Persons with obesity will be randomized to receive weight loss with or without supervised exercise. Metabolic phenotyping studies will be performed in both groups in the weight reduced state and compared to a group of obese persons not undergoing weight loss. All participants will be followed for a period of 1 year following metabolic phenotyping to track longitudinal changes in weight and other relevant outcomes measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Persons with obesity who do not undergo weight loss will participate in an inpatient assessment to measure metabolic responses to a 3 day eucaloric diet or a 3 day overfeeding challenge. Participants will be followed for 1 year after the metabolic studies to track longitudinal changes in body weight and other relevant health outcomes.
  Interventions: Other: Overfeeding
- Reduced obese + diet + exercise (Experimental): Persons with obesity randomized to a weight loss program consisting of caloric restriction, behavioral support, and supervised endurance exercise training. Following weight loss persons in this group will participate in an inpatient assessment to measure metabolic responses to a 3 day eucaloric diet or a 3 day overfeeding challenge. Participants will be followed for 1 year after the metabolic studies to track longitudinal changes in body weight and other relevant health outcomes.
  Interventions: Other: Weight Loss; Other: Exercise training; Other: Overfeeding
- Reduced obese + diet group (Active Comparator): Persons with obesity randomized to a weight loss program consisting of caloric restriction and behavioral support. Following weight loss persons in this group will participate in an inpatient assessment to measure metabolic responses to a 3 day eucaloric diet or a 3 day overfeeding challenge. Participants will be followed for 1 year after the metabolic studies to track longitudinal changes in body weight and other relevant health outcomes.
  Interventions: Other: Weight Loss; Other: Overfeeding

INTERVENTIONS:
Other: Weight Loss — 12-wk weight loss intervention using a meal replacement strategy (Health & Nutrition Technology, Carmel, CA), with an 8-10% weight loss goal
  Arms: Reduced obese + diet + exercise; Reduced obese + diet group
Other: Exercise training — 16-wk supervised endurance exercise training program
  Arms: Reduced obese + diet + exercise
Other: Overfeeding — 3-day hypercaloric diet designed to overfeed by 40% above total daily energy requirements

SUMMARY:
To more effectively address the problem of weight regain following weight loss for obese individuals, this study will evaluate the underlying biology of the reduced obese state. In depth studies of appetite, energy expenditure, physical activity levels and fat metabolism will be completed in obese and reduced obese individuals; with the latter subdivided into those who have lost weight with diet alone or diet plus exercise. Individuals will be studied following a brief overfeeding period to better understand how differences in biological responses to overeating might be involved in promoting or protecting against weight gain.

DETAILED DESCRIPTION:
The persistent problem of weight regain following weight loss is perhaps the most significant barrier to addressing the current obesity epidemic. The biological drive to regain weight following weight loss is due in part to increased appetite leading to increased energy intake (EI) and reductions in energy expenditure (EE) in part due to changes in energy expended in physical activity (PA). These physiological adaptations to weight loss are most relevant during episodes of dietary indiscretion resulting in overfeeding (OF) when reduced obese (RO) people fail to respond to the state of positive energy balance in a way that maintains the reduced state. There is increasing evidence that RO individuals who exercise (RO-Ex) are less like to regain as compared to RO individuals who are sedentary (RO-Sed). Previous studies were conducted on the effects of OF on EI, EE, PA and fat metabolism in non-obese individuals either prone (OP) or resistant to obesity (OR). Subjects were then followed for 5 years to measure weight change. These studies showed that differences in the response of nocturnal fat oxidation and higher levels of moderate/vigorous PA following OF correlated with 5 year weight gain suggesting that these factors were potentially important mechanisms for weight gain. Previous work has shown that measures of hunger fail to suppress with OF in RO individuals and that nocturnal fat oxidation is reduced in RO-Sed but maintained in RO-Ex following a day that included a bout of exercise. This study will look at the responses of EE, EI, PA and fat metabolism to OF (40% above basal energy for 3 days) in obese, RO-Sed and RO-Ex men and women and correlate these responses to weight change over the subsequent year. The hypothesis is that changes in the response of one or more of these variables to OF will correlate with weight regain. The Significance of the studies lies in the fact that subjects will begin to clarify the metabolic mechanisms that underlie a propensity for weight regain in RO individuals. Innovation: The proposed studies will systematically examine a range of responses to OF and prospectively correlate them with weight gain while taking into account aspects of behavior relevant to weight regain. The hope is that these studies will lay a foundation for future studies that will examine the mechanisms underlying specific adaptive responses that directly relate to weight regain and help with the design of strategies to address and/or respond to these processes.

ELIGIBILITY:
Inclusion criteria.

* BMI of 30-38 kg/m2 and weight stable over the previous 6 months.
* Satisfied with current weight and not planning to lose weight at the time of enrollment (persons with obesity control group) -or- not satisfied with current weight and motivated to lose weight at the time of enrollment (reduced obese groups)
* No more than 90 min or 3 bouts of planned physical activity/wk.
* Pass a medical and physical screening performed by the study physician.
* Reporting a habitual, regular sleep-wake cycle for the month preceding screening that involved going to bed between 2200 and 0100 h and getting up between 0600 and 0900 h with >7 h and <9.25 h in bed.
* Live or work within 45 minutes of the CU-AMC (reduced obese groups only) (exceptions may be made at the discretion of the Study PI on a case by case basis for highly motivated subjects).
* Own a smartphone (Android or Apple iOS).
* For Females
* Not currently pregnant or lactating
* Not pregnant within the past 6 months
* Not planning to become pregnant in the next 12 months; sexually active women of childbearing potential may be enrolled if they use a reliable means of contraception
* Capable and willing to provide informed consent, understand exclusion criteria, and accept the randomized group assignment (reduced obese groups)

Exclusion criteria.

* Being considered unsafe to participate as determined by the study physician;
* Taking medications affecting weight, triglycerides, or energy intake/energy expenditure in the last 3 months;
* Having abnormal blood chemistry and/or hematology as deemed significant by the study physician;
* Ever having a history of systemic, psychiatric, neurological disease, or drug and alcohol abuse;
* History of cardiovascular disease, diabetes, uncontrolled hypertension, untreated thyroid, renal, hepatic diseases, dyslipidemia or any other medical condition affecting weight or lipid metabolism;
* Score > 18 on Beck Depression Index (BDI) will require further assessment by the study physician to determine if it is appropriate for the subject to participate in the study;
* Use of a continuous positive airway pressure (CPAP) device for the treatment of obstructive sleep apnea (OSA). A score of >10 on the Epworth sleepiness scale or >5 on the Pittsburgh Sleep Quality Index will require further assessment by the study physician to determine if it is appropriate for the subject to participate in the study;
* Being positive for human immunodeficiency virus or hepatitis B or C;
* History of surgical procedure for weight loss at any time (e.g. gastroplasty, gastric bypass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve);
* Being a smoker or having been a smoker in the previous 6 months;
* Abnormal eating patterns identified by registered dietitian interview (dietary fat<15%, dietary fat>45%, dietary protein >30%);
* Working night shifts;
* Night eating syndrome (at least 25% of food intake is consumed after the evening meal and/or at least two episodes of nocturnal eating per week);
* Traveling > 2 time zones 2 weeks prior to an inpatient CTRC study visit;
* Currently participating in any formal weight loss or physical activity programs or clinical trials.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Fat oxidation as a correlate of weight regain as measured by room calorimetry | 24 hour period on day 7 of two diet conditions - one overfed & one eucaloric condition; weeks 16 & 20
  Fat oxidation as a correlate of weight regain will be assessed in both reduced obese groups with room calorimetry on two occasions, once after 3 days of overfeeding and once after 3 days of an energy balanced diet.

SECONDARY OUTCOMES:
Body weight per scale | Baseline, after 12 week weight loss intervention and 1 year after the end of second study condition
  Body weight will be measured via clinic scale. Change in body weight in response to the weight loss intervention
Body Composition via DXA | Baseline, after 12 week weight loss intervention and 1 year after the end of second study condition
  Body composition will be measured via DXA, Change in body composition in response to the weight loss intervention
Change in substrate utilization as measured by room calorimetry | 24 hour period, on day 7 of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and week 16 & 20 for reduced groups
  Substrate utilization will be measured by room calorimetry (change = overfeeding diet condition - eucaloric diet condition)
Change in nocturnal lipolysis as measured by use of stable isotope tracer | 24 hour period, on day 7 of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  Lipolysis will be measured using stable isotope tracers (change = overfeeding diet condition - eucaloric diet condition)
Change in total energy expenditure (TEE) as measured by room calorimetry | 24 hour period, on day 7 of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  TEE will be measured by room calorimetry (change = overfeeding diet condition - eucaloric diet condition)
Change in spontaneous physical activity (SPA) as measured by accelerometers | 7 days, on days 4-10 of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  SPA will be measured using accelerometers (change = overfeeding diet condition - eucaloric diet condition)
Change in spontaneous food intake measured with an ad libitum diet | 3 days - on days 8-10 - of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  Spontaneous food intake will be measured during a 3 day ad libitum diet (change = overfeeding diet condition - eucaloric diet condition)
Change in hunger and satiety using Visual Analog Scale | 3 days - on days 8-10 - of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  Hunger and satiety will be measured using visual analog scales (change = overfeeding diet condition - eucaloric diet condition)
Change in 24h hormone and metabolite profiles as measured by assay of plasma samples | 3 days - days 8-10 - of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  24h hormone and metabolite profiles will be assayed in plasma samples obtained during inpatient study visits (change = overfeeding diet condition - eucaloric diet condition)
Lipolysis as a correlate of weight regain as measured by stable isotope tracer | 24 period, on day 7 of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  Lipolysis as a correlate of weight regain will be assessed in both reduced obese groups with a stable isotope tracer on two occasions, once after 3 days of overfeeding and once after 3 days of an energy balanced diet.
Total energy expenditure (TEE) as a correlate of weight regain as measured by room calorimetry | 24 period, on day 7 of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  TEE as a correlate of weight regain will be assessed in both reduced obese groups with room calorimetry on two occasions, once after 3 days of overfeeding and once after 3 days of an energy balanced diet.
Spontaneous physical activity (SPA) as a correlate of weight regain as measured by accelerometers | 7 days, on days 4-10 of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  SPA as a correlate of weight regain will be assessed in both reduced obese groups with accelerometers on two occasions, once after 3 days of overfeeding and once after 3 days of an energy balanced diet.
Spontaneous food intake as a correlate of weight regain as measured with an ad libitum diet | 3 days - days 8-10 of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  SPA as a correlate of weight regain will be assessed in both reduced obese groups with an ad libitum diet on two occasions, once after 3 days of overfeeding and once after 3 days of an energy balanced diet.
24h hormone and metabolite profiles as a correlate of weight regain as measured by assay of plasma samples | 24 period, on day 7 of two diet conditions - eucaloric and overfed; week 1 and 4 for controls and weeks 16 and 20 for reduced
  24h hormone and metabolite profiles as a correlate of weight regain will be assessed in both reduced obese groups by assay of plasma samples on two occasions, once after 3 days of overfeeding and once after 3 days of an energy balanced diet.
Total daily energy expenditure as a correlate of weight regain as measured by doubly labeled water | two 1 week periods at 1 month and 1 year after second diet condition; week 8 and week 56 for controls and week 24 and week 72 for reduced
  Total daily energy expenditure as a correlate of weight regain will be measured in both reduced obese groups using doubly labeled water after the second diet condition intervention
Correlates of Weight Regain as measured by questionnaire | 30 minutes at baseline and every 8 weeks for 1 year following second diet condition; weeks 12, 20, 28, 36, 44, 52 for controls and weeks 28, 36, 44, 52, 60, 68, for reduced.
  Correlates of weight regain will be assessed in both reduced obese groups with questionnaires periodically over the intervention and follow-up period

OTHER OUTCOMES:
Change in fitness as measured by indirect calorimetry | 30 minutes at baseline and 1 year following second diet condition; Reduced group will have an additional measurement at week 12 following weight loss period.
  Fitness will be measured using indirect calorimetry during a graded exercise test to volitional exhaustion

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bessesen, MD, Principal Investigator — University of Colorado Anschutz Health and Wellness Center
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No